CLINICAL TRIAL: NCT03234738
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Intravenous TP-271 in Healthy Adult Subjects
Brief Title: A Phase 1 Safety and PK Study of IV TP-271
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: TP-271-002; HHSN272201100028C (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2017-07-06; First posted 2017-07-31 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — TP-271

STUDY DESIGN:
Intervention Model Description: Five Multiple-Ascending Doses
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: IV bags and lines are covered to prevent unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A (Active Comparator): Multiple IV doses of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 0.5 mg/kg once daily for 7 days, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271; Drug: Placebo
- Cohort B (Active Comparator): Multiple IV doses of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 1.0 mg/kg once daily for 7 days, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271; Drug: Placebo
- Cohort C (Active Comparator): Multiple IV doses of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 2.0 mg/kg once daily for 7 days, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271; Drug: Placebo
- Cohort D (Active Comparator): Multiple IV doses of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 2.5 mg/kg once daily for 7 days, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271; Drug: Placebo
- Cohort E (Active Comparator): Multiple IV doses of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 3.0 mg/kg once daily for 7 days, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271; Drug: Placebo

INTERVENTIONS:
Drug: TP-271 — multiple oral doses of TP-271 or placebo, dosed once daily for 7 days, randomized 3:1, doses escalating as 0.5 mg/kg, 1.0 mg/kg, 2.0 mg/kg, 2.5 mg/kg, and 3.0 mg/kg
Drug: Placebo — Placebo is sterile 0.45% saline randomized 3:1 to receive

SUMMARY:
This is a single-center, randomized, placebo-controlled, double-blind, multiple-ascending-dose, inpatient study to assess the safety, tolerability, and pharmacokinetics of TP-271 in healthy subjects. Subjects aged 18 to 50 years who fulfill the inclusion/exclusion criteria will be enrolled in this study.

DETAILED DESCRIPTION:
Up to 5 cohorts of 8 subjects each (up to a total of 40 subjects) will be enrolled. The 8 subjects within each cohort will be randomized 6:2 to receive multiple IV doses of TP-271 or placebo. Study drug will be administered IV once daily on the morning of Days 1 through 7 following an overnight fast (minimum 8 hours). The planned doses for study drug for Cohorts A - E are 0.5 mg/kg TP-271 or placebo, 1.0 mg/kg TP-271 or placebo, 2.0 mg/kg TP-271 or placebo, 2.5 mg/kg TP-271 or placebo and 3.0 mg/kg TP-271 or placebo respectively.

During the Screening period (Days -28 to -2 prior to the subject receiving TP-271 or placebo), each subject will be assessed for eligibility. Each subject must sign and date the ICF prior to undergoing any study-related procedures.

All cohorts will follow the same study design. On Day -1, subjects will be admitted to the study unit and eligibility confirmed. On Day 1, eligible subjects will be enrolled and randomized to receive either TP-271 or placebo and will receive the assigned drug from Days 1 through 7. Subjects will be required to stay at the study unit from Days -1 through 11 to assess safety and obtain the required PK samples. On Day 11, subjects will be discharged from the study unit. A final safety assessment will be performed once between Days 14 and 20, 7 to 13 days following administration of the subject's final dose of study drug.

After all 8 subjects in a cohort have completed study procedures through Day 11, the Principal Investigator and the Sponsor's Medical Monitor will evaluate all blinded safety and plasma PK data to determine whether any criteria that would require a meeting of the Safety Monitoring Committee (SMC) are met. If no such criteria are met, the study may proceed to the subsequent cohort at the next higher dose of TP-271 without consulting the SMC.

ELIGIBILITY:
Inclusion Criteria:

1. Be within the age range of 18 to 50 years, inclusive, at the time of Screening
2. Voluntarily sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved ICF to participate in the study after all relevant aspects of the study have been explained and discussed with the subject and before undergoing any study-related procedures
3. Have a body mass index (BMI) ≥18.0 and ≤33.0 kg/m2
4. Have a negative history of and negative screening results for human immunodeficiency virus 1 and 2 and hepatitis B and C antibodies
5. Have the ability to communicate with the study unit staff in a manner sufficient to carry out all protocol procedures as described
6. For female subjects, be of non-childbearing potential, either 1 year postmenopausal or surgically sterile (bilateral oophorectomy, bilateral tubal ligation, or complete hysterectomy)
7. For male subjects, be willing and able to use a barrier method of contraception or practice abstinence (including males who had a vasectomy) from dosing through 90 days after administration of the final dose of study drug

Exclusion Criteria:

1. History and/or presence of any clinically significant disease or disorder such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal, endocrine, psychiatric, or mental disease or disorder, or mental or legal incapacitation, which, in the opinion of the PI or Sub-Investigator(s), may either put the subject at risk because of participation in the study, influence the results of the study, or influence the subject's ability to participate in the study
2. Clinical laboratory values that fall outside the eligibility range specified in Appendix D; for laboratory values that are not included in Appendix D, values outside the reference range are exclusionary, with the following exceptions (Table 4. Acceptable Out-of-Range Clinical Laboratory Values
3. Known allergy to tetracycline antibiotics or to any of the excipients in TP-271
4. Clinically significant abnormality on a 12-lead ECG, including the following:

   * Rhythm other than sinus
   * Corrected QT interval using Fridericia's formula (QTcF) >450 msec
   * Evidence of second- or third-degree atrioventricular block
   * Pathological Q-waves (defined as Q-wave >40 msec or depth >0.4 to 0.5 mV)
   * Evidence of ventricular pre-excitation
   * Evidence of complete left bundle branch block (BBB), right BBB, or incomplete left BBB
   * Intraventricular conduction delay with QRS duration >120 msec
   * ST segment abnormalities, unless judged by the PI or Sub-Investigator(s) to be non pathologic
5. History of seizures
6. History within 3 years of a positive result on a urine screen for drugs of abuse or a positive result at Screening for any of the following drugs of abuse: tetrahydrocannabinols, cocaine, opioids, phencyclidines, amphetamine, benzodiazepine, and barbiturates
7. Use of tobacco, nicotine, or nicotine-replacement products within 3 months prior to administration of the study drug through the last visit
8. Typical weekly alcohol consumption of 7 or more alcoholic drinks, where 1 alcoholic drink is defined as 1 glass of beer (approximately 10 to 12 oz), 1 can (12 oz) of beer, 1 glass of wine (approximately 4 to 5 oz), or distilled spirits (approximately 1 oz or 30 mL of liquor)
9. Alcohol consumption within 48 hours prior to dosing
10. Participation in a clinical study within 10 half-lives of the prior study drug administration or within the previous 3 months if the half-life or dose of the investigational agent is unknown or planned participation in another clinical study concurrent with the current clinical study
11. History of difficulty donating blood or poor venous access
12. Blood donation (1 unit or approximately 350 mL) within 1 month prior to receiving study drug or plans to donate prior to receiving study drug or during the clinical study
13. Use of any prescription or nonprescription medication, including vitamins or herbal medications, vaccination, or immunization within 7 days or 5 half-lives (if known), whichever is longer, prior to dosing of study drug, with the following exceptions: medications used to treat an AE, and the use of acetaminophen, naproxen, and ibuprofen (except for within 24 hours prior to dosing)
14. Male subject donates or plans to donate sperm during the study and for at least 90 days after study drug administration.
15. Unwillingness or inability to follow the procedures outlined in the clinical study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Throughout the study, ~ 49 days
  Incidence, intensity, and type of adverse events (AEs) from the time of signing the informed consent form (ICF) through the EOS Visit
Physical Exams | ~ 20 days
  Changes in physical examination findings between Day -1 and the EOS Visit
Vital Signs | ~ 20 days
  Changes in vital signs from Day -1 through the EOS Visit
Safety Laboratory Results | ~ 20 days
  Changes in safety laboratory (clinical chemistry, electrolytes, hematology, blood glucose, and coagulation) results from Day -1 through the EOS Visit
ECG measurements | ~ 20 days
  Changes in electrocardiogram (ECG) measurements from Day -1 through the EOS Visit

SECONDARY OUTCOMES:
Assess the Pharmacokinetics (PK) of TP-271in Plasma | ~11 days
  Plasma concentrations of TP-271 and its C-4 epimer, TP-9555, for PK analysis from Days 1 through 11
Assess the Pharmacokinetics (PK) of TP-271 in Urine | ~11 days
  Urine concentrations of TP-271 and its C-4 epimer, TP-9555, from Days 1 through 11

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No